CLINICAL TRIAL: NCT03577704
Title: An Exploratory Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of HLX07 (Recombinant Anti-EGFR Humanized Monoclonal Antibody) Combined With Chemotherapy in Patients With Advanced Solid Tumors.
Brief Title: The Safety,Efficacy of Anti-EGFR Humanized Monoclonal Antibody Combined With Chemotherapy in Advanced Solid Tumors.
Acronym: HLX07Ib/II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-002
Record Dates: First submitted 2018-06-11; First posted 2018-07-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Gemcitabine; Cisplatin; Paclitaxel; Carboplatin; Oxaliplatin; Injections

STUDY DESIGN:
Intervention Model Description: The study used the Bayes optimal interval design (BOIN) to assign the subject's dose level and determine the maximum tolerated dose (MTD) of HLX07 in combination with chemotherapy.Each cohort contains 3 subjects and the patient in the first cohort receives treatment at the lowest dose level (single dose of 400 mg). The decision to increase or decrease the dose after each train is based on the probability of a predefined safety and toxicity threshold. When the observed rate of dose limiting toxicity (DLT) is less than 0.237 (low target safety margin), the dose for the next cohort escalates; when the observed rate of DLT is higher than 0.359 (target high toxicity cutoff), the dose deescalates. Otherwise, the dose remains the same. After each cohort is finished, a safety review committee will be held to determine the escalates or deescalates in the next cohort. The enrollment continues until the maximum 30 patients are reached.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HLX07+Gemcitabine+Cisplatin arm (Experimental): HLX07 is given on D1,D8,D15 combine with Gemcitabine (1000 mg/m2) and Cisplatin (75 mg/m2) in 3 weeks- cycles for 4-6 cycles .Gemcitabine was administered on the D1 and D8 and cisplatin 75 mg/m2 was administered on the D1. After 4-6 cycles of combination therapy, once weekly HLX07 infusion will be continue for a maximum duration of 2 years or until disease progression or emergence of intolerable toxicity or permanent withdrawal or death (whichever comes first).
  In each cohort, HLX07 will use BOIN design to assign the subject's dose level and determine the MTD.
  Interventions: Drug: HLX07+Gemcitabine+Cisplatin
- HLX07+Paclitaxel+Carboplatin arm (Experimental): HLX07 is given on D1,D8,D15 combine with Paclitaxel (80 mg/m2) and carboplatin (AUC=2) in 3 weeks-cycle for 4-6 cycles .Paclitaxel and carboplatin were administered on D1, D8 and D15. After 4-6 cycles of combination therapy, once weekly HLX07 infusion will be continue for a maximum duration of 2 years or until disease progression or emergence of intolerable toxicity or permanent withdrawal or death (whichever comes first).
  In each cohort, HLX07 will use BOIN design to assign the subject's dose level and determine the MTD.
  Interventions: Drug: HLX07+Paclitaxel+Carboplatin
- HLX07+mFOLFOX6 arm (Experimental): HLX07 is given on D1,D8 combine with mFOLFOX6 ( oxaliplatin (85 mg/m2), leucovorin (400 mg/m2), and 5-FU (400 mg/m2, followed by 2400 mg/m2) in 2 weeks-cycles for 6-12 cycles . Oxaliplatin, leucovorin and 5-FU were administered on D1. After 6-12 cycles of combination therapy,once weekly HLX07 infusion will be continue for a maximum duration of 2 years or until disease progression or emergence of intolerable toxicity or permanent withdrawal or death (whichever comes first).
  In each cohort, HLX07 will use BOIN design to assign the subject's dose level and determine the MTD.
  Interventions: Drug: HLX07+mFOLFOX6

INTERVENTIONS:
Drug: HLX07+Gemcitabine+Cisplatin — Recombinant anti-EGFR humanized monoclonal antibody in combination with Gemcitabine and Cisplatin.
  HLX07, IV, weekly.
  Other Names: Recombinant anti-EGFR humanized monoclonal antibody; Gemzar; Cisplatin
  Arms: HLX07+Gemcitabine+Cisplatin arm
Drug: HLX07+Paclitaxel+Carboplatin — Recombinant anti-EGFR humanized monoclonal antibody in combination with Paclitaxel and Carboplatin.
  HLX07, IV, weekly.
  Other Names: Recombinant anti-EGFR humanized monoclonal antibody; Paclitaxel; Carboplatin
  Arms: HLX07+Paclitaxel+Carboplatin arm
Drug: HLX07+mFOLFOX6 — Recombinant anti-EGFR humanized monoclonal antibody in combination with Oxaliplatin, Calcium Folinate and 5-FU.
  HLX07, IV, weekly.
  Other Names: Recombinant anti-EGFR humanized monoclonal antibody; Oxaliplatin for Injection; Folinic acid calcium salt hydrate; 5-fluouracil
  Arms: HLX07+mFOLFOX6 arm

SUMMARY:
HLX07 is a new anti-EGFR monoclonal antibody (mAb) with improved glycosylation pattern.In pre-clinical efficacy studies, HLX-07 is either equivalent or more potent than cetuximab in multiple cancer models without increased toxicities.This study is an open-labeled, dose-escalation study designed to explore the maximum tolerated dose (MTD) and safety of HLX07 in combination with different chemotherapy regimens.

DETAILED DESCRIPTION:
This study is a parallel 3-arm escalation trial with 3 doses of HLX07 (400 mg, 600 mg, or 800 mg per single dose) combined with 3 different fixed-dose chemotherapy regimens.

Three chemotherapy regimens are：

① Gemcitabine (1000 mg/m2) and Cisplatin (75 mg/m2) , every three weeks. Gemcitabine was administered on the first day and on the 8th day, and cisplatin 75 mg/m2 was administered on the first day , a total of 4-6 cycles。

② Paclitaxel (80 mg/m2) and carboplatin (AUC=2), every 3 weeks. Paclitaxel and carboplatin were administered on days 1, 8 and 15 for a total of 4-6 cycles.

③ mFOLFOX6 protocol: oxaliplatin (85 mg/m2), leucovorin (400 mg/m2), and 5-fluouracil (5-FU) (400 mg/m2, followed by 2400 mg/m2), every 2 weeks. Oxaliplatin, leucovorin and 5-FU were administered on the first day.

After 4 to 6 cycles of (gemcitabine and cisplatin regimens) and (the paclitaxel and carboplatin regimens) or after 6 to 12 cycles of the mFOLFOX6 regimen, well-controlled patients will be continue to receive a weekly HLX07 infusion as maintenance therapy for maximum 2 years or until disease progression or emergence of intolerable toxicity or permanent withdrawal or death (whichever comes first).

The study used the Bayes optimal interval design (BOIN) to determine the MTD of HLX07 in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed metastatic or recurrent advanced solid tumors which has indication to receive treatment with one of above three chemotherapy regimens.The lesions must be assessable based on the RECIST v1.1 criteria.The number of previously received chemotherapy regimens should not exceed two.
2. At least 28 days from prior major surgery, prior cytotoxic chemotherapy, or prior therapy with investigational agents or local radiotherapy and at least 42 days from the last infusion of immune check point inhibitors (The antibodies or drugs include but not limited to IDO, PD-1, PD-L1, IL-2R, CTLA-4, CD137, and GITR) before the first infusion of investigational product.
3. Eastern Cooperative Oncology Group (ECOG) score ≤ 1,
4. Expected survival time ≥ 3 months;
5. Has sufficient hematological function, defined as: neutrophil absolute value ≥ 1.5 × 109 / L; hemoglobin level ≥ 9.0 g / dL ; Platelet count ≥100×109 /L.
6. Has sufficient liver function, defined as: total bilirubin level ≤ 1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN, For patients with known liver metastases or primary hepatocellular carcinoma patients ≤ 5 x ULN.
7. Has adequate coagulation function defined as: International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 x ULN, and activated partial thromboplastin time (PTT) in the absence of anticoagulant therapy /aPTT) ≤ 1.5 x ULN.
8. Has adequate cardiac function, defined as: left ventricular ejection fraction (LVEF) ≥ 50%.
9. Has sufficient renal function; in patients receiving the gemcitabine plus cisplatin regimen is defined as creatinine clearance ≥ 60 ml/min and in patients receiving the paclitaxel plus carboplatin regimen or the mFOLFOX6 regimen, is defined as creatinine clearance ≥ 50 ml/min (calculated by the Cockcroft-Gault formula).
10. Use of effective contraceptive measures if procreative potential exists.
11. Able to provide written informed consent.

Exclusion Criteria:

1. Concurrent unstable or uncontrolled medical conditions. Either of the followings:

   * Active systemic infections;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg), or poor compliance with anti-hypertensive agents;
   * Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association (NYHA)) or acute myocardial infarction within 6 months;
   * Uncontrolled diabetes or poor compliance with hypoglycemic agents;
   * The presence of chronically unhealed wound or ulcers;
   * Other chronic diseases, which, in the opinion of the investigator, could compromise safety of the patient or the integrity of study.
2. Unstable central nervous system (CNS) metastasis. Patients who have previously undergone surgery or radiotherapy for brain metastases may participate in this study if they are clinically stable for at least 4 weeks and has stopped steroids for at least 2 weeks prior to the first infusion of the test drug and there is no new evidence of progression.
3. Has primary central nervous system malignancy;
4. Known patients have drug allergies to specific drug regimens (eg anti-EGFR monoclonal antibodies, gemcitabine, platinum, paclitaxel, fluorouracil allergy);
5. known active hepatitis B or C infection (active hepatitis B is defined as hepatitis B surface antigen HBsAg positive and Hepatitis B virus (HBV) DNA> 500 copies / ml; active hepatitis C is defined as hepatitis C antibody-positive and / or quantitative Hepatitis C virus (HCV) RNA results positive);
6. Human immunodeficiency virus infection .
7. Pregnancy or breast-feeding woman.
8. Patients with colorectal cancer whose tumors have K-ras, N-ras, or B-raf mutations;
9. The patient has a history of alcohol abuse or drug abuse;
10. Use of herbal medicine within the first 2 weeks before the first infusion of the test drug;
11. Treatment with systemic steroids (equivalent to >10 mg/day of methylprednisolone) or any other form of immunosuppressive therapy within 2 weeks of the first infusion of the test drug;
12. Patient has a history or current evidence of any condition or disease that could confound the results of the study, or is not the best interest of the patient to participate, in the opinion of Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of HLX07 combined with different chemotherapy regimen | up to 24 months
  The incidence of DLT combined with different chemotherapy regimens based on NCI CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Jin E Li, PhD, Principal Investigator — No.1800 Yuntai Road,Pudong District,Shanghai
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] M.M. Hou, C.L. Ho, H.Y. Lin, W. Jiang, S. Liu, Y. Hong, A. Luk, S.F. Lin, T.C. Hsieh, E. Liu. A novel anti-EGFR antibody HLX07 for potential treatment of squamous cell carcinoma of the head and neck. Annals of Oncology. Volume 30 | Supplement 9 | November 2019.
- See also: ESMO Asia 2019 (Poster); Annals of Oncology — https://doi.org/10.1093/annonc/mdz420.007